CLINICAL TRIAL: NCT00698711
Title: Vaccination of Prostate Cancer Patients With MUC-2-KLH Conjugate Plus the Immunological Adjuvant QS21: A Trial Comparing MUC-2-KLH Doses
Brief Title: Vaccination of Prostate Cancer Patients With MUC-2-KLH Conjugate Plus the Immunological Adjuvant QS21
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-122
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; MUC-2-KLH; QS 21
MeSH Terms: conditions — Prostatic Neoplasms | interventions — MUC-2-KLH vaccine

ARMS (1):
- 1 (Experimental): Three groups of 5 patients enrolled sequentially comprised from will receive MUC-2-KLH vaccines at the following g amounts of MUC-2-KLH per vaccination.
  10 + 100 μg QS21 30 + 100 μg QS21 3 + 100 μg QS21
  Interventions: Biological: MUC-2-KLH

INTERVENTIONS:
Biological: MUC-2-KLH — The MUC-2-KLH conjugate will be administered subcutaneously to random sites on the upper arm and upper leg at weekly intervals for 3 weeks. This will be followed by a 4 week break and then a fourth vaccination during week 7, and 3 months later during week 19. Booster vaccinations may be given at or after week 50 and 100, and every 6 months thereafter to select patients who show no evidence of radiographic disease progression.
  After 5 patients have been enrolled and completed two vaccinations without Grade II or greater toxicity, we will proceed to the next higher dose level. No dose escalations will be performed in the same patient.

SUMMARY:
The purpose of this research is to help us study a vaccine treatment for patients with prostate cancer. A vaccine is a medicine that teaches the body to destroy harmful infections and other foreign substances. The immune system is made up of many different types of cells, which fight infection and disease in your body. A vaccine may stimulate the immune system to destroy the cancer cells. It may also help to slow the growth of the cancer. The vaccine is a solution given as an injection given into or under the skin. It is made up of several parts. The first part is MUC-2, a protein present in many cancers, especially prostate cancer. MUC-2 is attached to a material called KLH or keyhole limpet hemocyanin. KLH is purified from a snail- like marine mollusk called a keyhole limpet and has been used for many years to boost immune responses in animals and in people. Attaching MUC-2 to KLH helps the immune system react to MUC-2. The mixture of MUC-2 attached to KLH is in turn mixed with a material called QS21, from the bark of a tree, which also helps the immune system to make more cancer- fighting cells. A vaccine like the one you will receive has been given to laboratory animals and been shown to produce an immune response in these animals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate cancer that is histologically confirmed by the Department of Pathology at MSKCC will be considered if they show progression of disease based on biochemical parameters. Patients with radiographic evidence of disease are not eligible.
* Hormonal status will be recorded on the basis of serum testosterone levels.
* Patients who have progressed after primary therapy to include surgery or radiation (with or without neo-adjuvant androgen ablation), or intermittent hormonal treatment who have non-castrate levels of testosterone (>50 ng/ml). Patients with soft tissue and/or bone disease or patients who are androgen- independent with no evidence of radiographic disease are not eligible. Those patients who are symptomatic or who are anticipated to develop symptoms within 6 months of entry will be excluded.
* Patients should have no change in their hormone therapies (with the exception of therapies needed to maintain castrate levels of testosterone), including prednisone or dexamethasone within two weeks prior to entry into study.
* Patients must have evaluable disease (by serial changes in PSA).
* Karnofsky performance status >60%.
* Patients must have adequate organ function as defined by:
* WBC > or = to 3500/mm3 platelet count > or = to 100,000 mm3.
* Bilirubin < or = 2.0 rag/100 ml or SGOT <3.0 X's the upper limit of normal.
* Creatinine < or = 2.0 mg/100 ml or creatinine clearance > or = 40 cc/min.
* Patients must have recovered from the toxicity of any prior therapy, and not received chemotherapy or radiation therapy for at least 4 weeks prior to entry into the trial.
* No history of an active secondary malignancy within the prior five years except for nonmelanoma skin cancer.
* Patients must be at least 18 years of age.
* Patients who have previously received suramin, may be treated if they have been off this drug for at least 8 weeks and/or ha ve a documented plasma concentration below 50 mg/ml. For these patients, replacement doses of hydrocortisone are permitted.
* Patients must sign informed consent.
* Registration to IRB Protocol 90-40 (Correlative studies in human prostate cancer).

Exclusion Criteria:

* Clinically significant cardiac disease (New York Heart Association Class III/IV), or severe debilitating pulmonary disease.
* Active CNS or epidural tumor.
* An infection requiring antibiotic treatment.
* Narcotic dependent pain.
* Anticipated survival of less than 6 months.
* Positive stool guaiac excluding hemorrhoids or history of documented radiation induced proctitis.
* Allergy to seafood.
* Patients with radiographic evidence of metastatic disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1997-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine an optimal dose of the MUC-2-KLH conjugate plus the immunological adjuvant QS21 in patient with prostate cancer that Induces an antibody response to MUC-2. and induces helper T and/or cytotoxic T cell response against MUC -2. | conclusion of study
To determine the safety of immunization with MUC-2-KLH conjugate prepared using an MBS heterobifunctional linker plus QS21. | conclusion of study
To determine the effect of MUC-2-KLH dose on the T cell response against MUC-2 and by skin testing. | conclusion of study

SECONDARY OUTCOMES:
To assess post-immunization changes in prostate specific antigen levels and other objective parameters or disease (radionuclide bone scan and/or measurable disease if present). | conclusion of study
To monitor changes in serum CASA levels prior to and following treatment. | conclusion of study
To monitor sequentially, the peripheral blood for the presence of PSA mRNA in circulating cells using a PCR based assay. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org